CLINICAL TRIAL: NCT03389126
Title: Phase II Study of Avelumab in Patients With Advanced Hepatocellular Carcinoma After Prior Sorafenib Treatment
Acronym: AvelumabHCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Kyung-Hun Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1708-040-876
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab 10 mg/kg every 2 wks until disease progression or unacceptable toxicity
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/kg intravenous injection every 2 weeks until disease progression or unacceptable toxicity
  Other Names: Bavencio

SUMMARY:
An open label, single arm, Phase II study of avelumab in patients with advanced hepatocellular carcinoma after prior sorafenib treatment

DETAILED DESCRIPTION:
This is an open label study of avelumab monotherapy. Patients with advanced hepatocellular carcinoma after prior sorafenib treatment are eligible. Patients should have failed to sorafenib or be intolerant to sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose of the study, provide signed and dated informed consent, and able to comply with all procedures
2. Male or female subjects aged ≥ 18 years
3. Histologically or cytologically proven advanced hepatocellular carcinoma not eligible for surgical and/or locoregional therapies; or progressive disease after surgical and /or locoregional therapies.
4. Patients who were intolerant to sorafenib or for whom sorafenib failed.
5. At least one RECIST 1.1 measurable untreated lesion. All subjects must have at least one previously untreated, unidimensionally measurable lesion by contrast-enhanced spiral computed tomography (CT) ≥ 10 mm or contrast enhanced dynamic magnetic resonance imaging (MRI) scan ≥ 10 mm (malignant lymph nodes must be ≥ 15 mm on short axis)
6. ECOG performance status of 0 to 1 at trial entry
7. Child-Pugh Class A
8. Subjects are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

   i) HBV-HCC: Resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or Chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA < 100 IU/mL and must be on antiviral therapy.

   ii) HCV-HCC: Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody
9. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test. Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists.
10. Males who are sexually active with WOCBP must agree to follow instructions for method of contraception as indicated in the informed consent form, for the duration of treatment with study drug plus 5 half-lives of the study drug plus 90 days.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. Prior liver transplant
3. Active, known, or suspected autoimmune disease
4. Pregnancy or lactation period
5. Participation in another clinical trial within the past 30 days
6. Inadequate hepatic function defined by a total bilirubin level > 3.0 mg/dl, an AST level > 5 × the upper limit of normal range (ULN), and an ALT level > 5 × ULN.
7. Inadequate renal function defined by an estimated creatinine clearance < 50 mL/min according to the Cockcroft-Gault formula or by measure of creatinine clearance from 24 hour urine collection
8. Inadequate hematologic function defined by WBC < 2000/μL, Platelets < 60,000/μL, Hemoglobin < 8.5 g/dL.
9. Active brain metastases or leptomeningeal metastases, requiring immunosuppressive doses of corticosteroids (> 10 mg/day prednisone equivalents).
10. IMMUNOSUPRESSANTS: "Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
11. AUTOIMMUNE DISEASE: "Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible."
12. ORGAN TRANSPLANTATION: "Prior organ transplantation including allogenic stem-cell transplantation."
13. INFECTIONS: "Active infection requiring systemic therapy. "
14. HIV/AIDS: "Known history of testing positive for HIV or known acquired immunodeficiency syndrome."
15. VACCINATION: "Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines "
16. HYPERSENSITIIVTY TO STUDY DRUG: "Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)"
17. CARDIOVASCULAR DISEASE: "Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication."
18. OTHER PERSISTING TOXICITIES: "Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable."
19. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
20. Any history of clinically meaningful variceal bleeding within the last three months 21, Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies (or other agents specifically targeting immune checkpoint pathway)

22. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
response rate | 6 weeks
  RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hun Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Data sharing should be decided upon formal documented requests.

REFERENCES:
- [Derived] Lee DW, Cho EJ, Lee JH, Yu SJ, Kim YJ, Yoon JH, Kim TY, Han SW, Oh DY, Im SA, Kim TY, Lee Y, Kim H, Lee KH. Phase II Study of Avelumab in Patients with Advanced Hepatocellular Carcinoma Previously Treated with Sorafenib. Clin Cancer Res. 2021 Feb 1;27(3):713-718. doi: 10.1158/1078-0432.CCR-20-3094. Epub 2020 Nov 2. PMID 33139266